CLINICAL TRIAL: NCT01851889
Title: Optimizing Continuous-flow Left Ventricular Assist Device Settings and Identification of Pump Malfunction - A Comparative Study of Echocardiography and Invasive Hemodynamics
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Finn Gustafsson, DMSc, Ph.d., Chief Physician., Rigshospitalet, Denmark
Other Study IDs: H-3-2013-010
Record Dates: First submitted 2013-04-29; First posted 2013-05-13 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Heart Failure.
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- CF-LVAD pump speed.

SUMMARY:
The purpose of the trial is to identify factors which can be used as guidance when optimizing continuous-flow left ventricular assist device (CF-LVAD) settings.

The hypothesis of the study is that pulmonary capillary wedge pressure (PCWP) will change independently of left ventricular end diastolic diameter (LVEDD) when increasing pump speed ie ΔPCWP/RPM ≠ ΔLVEDD/RPM.

The primary combined endpoint of the study is correlation between ΔPCWP and LVEDD slope under ramp testing in a cohort of "continuous-flow left ventricular assist device" heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure patients with HeartMate II (HM II) followed as outpatients at The Heart Centre at University Hospital of Copenhagen, Rigshospitalet.
* Age > 18 years.
* Heart failure in stable phase without the need for intravenous inotropic therapy.
* Ischemic or non-ischemic cardiomyopathy.
* Signed informed consent.

Exclusion Criteria:

* Unstable patients with the need for intravenous inotropic therapy.
* Current hospitalization.
* Implantation of HM II less than one month ago.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All heart failure patients with CF-LVAD at University Hospital of Copenhagen, Rigshospitalet.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Pulmonary capillary wedge pressure in mmHg. | On trial day.

CONTACTS AND LOCATIONS:
Overall Officials: Mette H Jung, MD, Principal Investigator — Department of Cardiology B, University Hospital Rigshospitalet.; Finn Gustafsson, MD, DMSc, PhD, Principal Investigator — Department of Cardiology B, University Hospital Rigshospitalet.
Locations (1):
- University Hospital Rigshospitalet., Copenhagen, Kbh Oe, Denmark